CLINICAL TRIAL: NCT05599256
Title: A Prospective, Single-arm Clinical Trial of Prevention of Severe Acute Graft-versus-host Disease After Pediatric Patients Receiving Allogeneic Hematopoietic Stem Cell Transplantation Using a daGOAT Model
Brief Title: Prevention of Severe Acute Graft-versus-host Disease in Pediatric Patients Using a daGOAT Model
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IIT2022034（child）
Record Dates: First submitted 2022-10-20; First posted 2022-10-31 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-03

CONDITIONS: Transplant-Related Disorder
MeSH Terms: interventions — ruxolitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The group of daGOAT model prevention (Experimental): Model-predicted high-risk patients: weight ≤ 25 kg, ruxolitinib, 2.5mg bid po until at least day 60 post-transplant and terminated after day 100; weight > 25 kg, ruxolitinib, 5mg bid po until at least day 60 post-transplant and terminated after day 100. If 'azoles' are taken concomitantly, ruxolitinib will start at half dose. If the patient tolerates ruxolitinib, the dose can be increased to 10mg bid po.
  Model-predicted low risk: regular aGVHD prophylactic regimens.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Model-predicted high-risk patients: weight ≤ 25 kg, ruxolitinib, 2.5mg bid po until at least day 60 post-transplant and terminated after day 100; weight > 25 kg, ruxolitinib, 5mg bid po until at least day 60 post-transplant and terminated after day 100. If 'azoles' are taken concomitantly, ruxolitinib will start at half dose. If the patient tolerates ruxolitinib, the dose can be increased to 10mg bid po.
  Model-predicted low risk: regular aGVHD prophylactic regimens.

SUMMARY:
To evaluate the efficacy and safety of ruxolitinib for prophylactic therapy of child patients who are predicted to have a high risk for developing severe acute graftversus-host disease (aGVHD) by the dynamic aGVHD Onset Anticipation Tianjin (daGOAT) model.

DETAILED DESCRIPTION:
This study aims to prospectively evaluate the use of the daGOAT model in real-world clinical settings at the Institute of Hematology, Chinese Academy of Medical Sciences (IHCAMS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≤ 16 years of age;
2. Patients receiving human leukocyte antigen mismatched and non-cord blood allogeneic hematopoietic stem cell transplantation;
3. Patients who can take oral medication;
4. Patients or their guardians have to sign an informed consent form before the start of the research procedure.

Exclusion Criteria:

1. Tandem transplantation or multiple transplantations;
2. Patients who are allergic to or cannot tolerate ruxolitinib;
3. Mental or other medical conditions that make the patients unable to comply with the research treatment and monitoring requirements;
4. Patients who are pregnant or cannot take appropriate contraceptive measures during treatment;
5. Patients who are ineligible for the study due to other factors, or will bear great risk if participating in the study.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Severe aGVHD during 100 days after transplantation according to the MAGIC criteria | 100 days after transplantation
  Incidence of severe aGVHD after transplantation within 100 days. The medical records for each case wil be reviewed by two or three physicians to confirm the aGVHD diagnosis and grading (according to the MAGIC criteria).

SECONDARY OUTCOMES:
aGVHD in various target organs during 100 days after transplantation according to the MAGIC criteria | 100 days after transplantation
  Incidence of aGVHD (any grade) in various target organs. The medical records for each case wil be reviewed by two or three physicians to confirm the aGVHD diagnosis and grading (according to the MAGIC criteria).
Overall survival during 1.5 year after transplantation | Days 14, 28, 42, 60, 90, 180, 270, 360 and 540 after transplantation
  Patients will be followed up at days 14, 28, 42, 60, 90, 180, 270, 360 and 540 after transplantation; data on survival will be collected.
Relapse-free survival rate and relapse rate during 1.5 year after transplantation | Days 14, 28, 42, 60, 90, 180, 270, 360 and 540 after transplantation
  Patients will be followed up at days 14, 28, 42, 60, 90, 180, 270, 360 and 540 after transplantation; data on relapse will be collected.
Incidence of infections during 1.5 year after transplantation | 1.5 year after transplantation
  Infection was defined as meeting one of the following criteria: culture-confirmed presence of bacteria or fungi in a sample collected from a sterile site; polymerase chain reaction-confirmed viremia at ≥ 5000 copies/ml for the cytomegalovirus or ≥ 10000 copies/ml for the Epstein-Barr virus; or body temperature ≥ 38 ℃ with culture-confirmed presence of pathogens from a non-sterile site.
Safety of treatment during 100 days after transplantation according to the Common Terminology Criteria for Adverse Events version 5.0 | 100 days after transplantation
  Data on adverse events of treatment will be collected.
Total cost of treatment during 1.5 year after transplantation | 1.5 year after transplantation
  Data on total cost of treatment will be collected from the medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

DOCUMENTS (1):
  • Study Protocol (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT05599256/Prot_002.pdf